CLINICAL TRIAL: NCT00512681
Title: A Phase II Study of S-1 Combined With Irinotecan and Oxaliplatin in Recurrent or Metastatic Gastric Carcinoma
Brief Title: A Phase II Study of Irinotecan, Oxaliplatin, Plus TS-1 in Untreated Metastatic Gastric Cancer
Acronym: TIROX2
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: National Cancer Center, Korea (Other Government)
Responsible Party: Sook Ryun Park, M.D, National Cancer Center, Korea
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: NCCCTS-07-264
Record Dates: First submitted 2007-08-07; First posted 2007-08-08 (Estimated); Last update posted 2009-09-18 (Estimated); Status verified 2009-09

CONDITIONS: Stomach Neoplasms
Keywords: Stomach Neoplasms; Secondary; Combination chemotherapy; S-1; irinotecan; oxaliplatin
MeSH Terms: conditions — Stomach Neoplasms; Neoplasm Metastasis | interventions — Irinotecan; Oxaliplatin; titanium silicide

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

INTERVENTIONS:
Drug: Irinotecan, Oxaliplatin, TS-1 — * S-1 40 mg/m2/day every 12-h p.o. on days 1(evening)-15 (morning)
  * Irinotecan 150 mg/m2 mixed in d5w 500 ml iv over 90-min on days 1
  * Oxaliplatin 85 mg/m2 mixed in d5w 250 ml iv over 2-h on days 1

SUMMARY:
Patients will be treated with irinotecan (150mg/m2) followed by oxaliplatin (85mg/m2)on day 1 and S-1(80mg/m2/day) from day 1 to 14 every 3 weeks. Patients will receive up to a planned treatment of maximum 12 cycles of chemotherapy. Response assessement will be performed every 2 cycles of chemotherapy.

ELIGIBILITY:
Inclusion Criteria:

1. Histologically or cytologically confirmed gastric adenocarcinoma with recurrent or metastatic disease
2. Age ≥18 years
3. Eastern Cooperative Oncology Group (ECOG) performance status 0-2
4. Disease status must be that of measurable disease as defined by RECIST criteria:Measurable lesions: Lesions that can be accurately measured in at least one dimension by any of the following: - CT of abdomen, pelvis or thorax, if the longest diameter to be recorded is at least 10 mm with spiral CT- Chest x-ray, if the lung lesion to be recorded is clearly defined and surrounded by aerated lung and the diameter to be recorded is at least 20 mm- Physical examination, if the clinically detected lesions are superficial (e.g., skin nodule and palpable lymph nodes) and at least 10 mm
5. No prior treatment for recurrent or metastatic disease; prior adjuvant/neoadjuvant therapy is allowed if at least 12 months have elapsed between completion of adjuvant/neoadjuvant therapy and enrolment into the study. However, prior oxaliplatin and/or irinotecan as adjuvant therapy are not allowed.
6. Adequate major organ function including the following: Hematopoietic function: ANC ³ 1,500/mm3, Platelet ³ 100,000/mm3Hepatic function: serum bilirubin 1.5 mg/dl, AST/ALT levels 2.5 x UNL ( 5 x UNL if liver metastases are present)Renal function: serum creatinine UNL
7. Patients should sign a written informed consent before study entry

Exclusion Criteria:

1. Prior history of peripheral neuropathy
2. Inadequate cardiovascular function:New York Heart Association class III or IV heart diseaseUnstable angina or myocardial infarction within the past 6 monthsHistory of significant ventricular arrhythmia requiring medication with antiarrhythmics or significant conduction system abnormality
3. Serious concurrent infection or nonmalignant illness that is uncontrolled or whose control may be jeopardized by complications of study therapy
4. Other malignancy within the past 3 years except non-melanomatous skin cancer or carcinoma in situ of the cervix
5. Psychiatric disorder that would preclude compliance
6. Pregnant, nursing women or patients with reproductive potential without contraception
7. Patients receiving a concomitant treatment with drugs interacting with S-1 such as flucytosine

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 44 (Estimated)
Dates: Start 2007-07; Primary Completion 2009-07 (Actual); Study Completion 2009-07 (Actual)

PRIMARY OUTCOMES:
Maximal overall response rate | During chemotherapy

SECONDARY OUTCOMES:
Progression-free survival,Overall survival,Toxicity assessment,&genetic polymorphism and association with chemical outcomes | during study period

CONTACTS AND LOCATIONS:
Overall Officials: Sook Ryun Park, M.D., Principal Investigator — National Cancer Center, Korea
Locations (1):
- National Cancer Center Korea, Goyang-si, Gyeonggi-do, South Korea